CLINICAL TRIAL: NCT05074407
Title: Neck Pain in Office Workers and Remote Workers During Covid 19 Pandemic
Brief Title: Neck Pain in Office Workers During Covid 19 Pandemic
Status: Completed | Type: Observational
Sponsor: Kırklareli University (Other)
Responsible Party: Principal Investigator, Betül Çiftçi Tepeli, dr, Kırklareli University
Other Study IDs: E-69456409-199-4707
Record Dates: First submitted 2021-10-06; First posted 2021-10-12 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Neck Pain
Keywords: neck pain; posture
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Work content of office workers are using computers, conferences, presentations and talking on the phones. Static postures and repetitive writing and reading activities at inappropriate body postures are the most common activities of office workers. Decreased physical activity and prolonged computer use cause occupational safety problems and musculoskeletal problems. Neck pain is one of the most common problem in office workers and the studies have shown the incidence of neck pain in office workers is 34-49% .

The aim of this study to evaluate the effects of remote employee in neck pain in Office workers during covid 19 pandemic

DETAILED DESCRIPTION:
The data of study was obtained by using online questionnaire. The questionnaire was generated through Google forms and the online questionnaire link was delivered via e-mail to office workers. The questionnaire link was active within 3 months for data collection. The information about study was stated and before answering the questionnaire, all participants were asked whether they were willing to participate in the study and thus all participants have declared voluntary for the study. All participants were employees such as clerical or administrative work in an office. The inclusion criteria were as follows; (a) being an office worker or remote employee; (b) aged between 18 and 55 years; (c). had a diagnosis with myofascial pain in neck. The exclusion criteria were as follows: (a) having a history of surgery in neck region; (b): a diagnosis with skeletal muscle diseases, chronic kidney diseases, chronic liver failure, malignancy and neurologic diseases; (c): having cognitive impairment that affects answering the online questionnaire properly; (d): having internet access and not being able to complete the online questionnaire; (e): being pregnant. The Beck Depression Inventory (BDI), The Nottingham Health Profile (NHP), Neck Pain and Disability Scale (NPDS), Pittsburgh Sleep Quality Index (PSQI), The Nottingham Health Profile (NHP) and demographic form were obtained

ELIGIBILITY:
Inclusion Criteria:

being an office worker or remote employee aged between 18 and 55 years had a diagnosis with myofascial pain in neck.

Exclusion Criteria:

* having a history of surgery in neck region a diagnosis with skeletal muscle diseases, chronic kidney diseases, chronic liver failure, malignancy and neurologic diseases having cognitive impairment that affects answering the online questionnaire properly having internet access and not being able to complete the online questionnaire being pregnant

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: office workers
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
The Beck Depression Inventory (BDI) | questionnaire takes five minutes
  The BDI has 21 items that describe symptoms of depression. The questionnaire is in a multiple-choice format, and each item has a four-point scale variable from 0 (absent) to 3 (severe). The minimum score is 0 and the maximum score is 63
The Nottingham Health Profile (NHP) | questionnaire takes five minutes
  The NHP has two parts. The first part of the NHP has six domains that include pain, emotional reaction, sleep, social isolation, physical abilities, and energy level. The second part of the NHP assesses the presence of difficulties with performing daily activities
Neck Pain and Disability Scale (NPDS) | questionnaire takes five minutes
  The NPDS contains 20 items related with 4 dimensions as neck problems, pain intensitiy, emotion-cognition and interference with life activities. Each item is a 100 mm VAS with 6 sections from 0 to 5 marked at equal intervals. The score of items is ranging 0 (no pain or activity limitation) and 5 ( much pain or maximal limitation ). activities. the range of total score is 0 to100 and higher score indicate greater disability.
Pittsburgh Sleep Quality Index (PSQI) | questionnaire takes five minutes
  The PSQI consists of 24 questions to assess patients'sleep dysfunction. 19 questions about sleep duration, latency and the frequency and severity of specific sleep-related problems. 5 questions are answered by the patient's bed partner or roommate and these five questions are used for clinical purposes. PSQI has seven components and the components are added to get global PSQI score. The global score has a range 0-21 and higher scores show lower sleep quality
demographic form | questionnaire takes five minutes
  Sociodemographic features including age, gender, marital status, education level, comorbid diseases, height, weight, kind of working (office worker or remote employee) were assessed.

CONTACTS AND LOCATIONS:
Overall Officials: betül çiftçi, Principal Investigator — Kırklareli University
Locations (1):
- Kırklareli University, Kırklareli, Turkey (Türkiye)

REFERENCES:
- [Derived] Ciftci B, Demirhan F. Investigating the impacts of working at home among office workers with neck pain on health status, depression and sleep quality during the COVID-19 pandemic. Int J Occup Saf Ergon. 2023 Sep;29(3):970-978. doi: 10.1080/10803548.2022.2090132. Epub 2022 Aug 9. PMID 35713149